CLINICAL TRIAL: NCT03542019
Title: The Endocrown; a Prospective Randomised Clinical Trial of Three Different Ceramics
Brief Title: Survival of Endocrowns Made From Different Ceramics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Ahmad El-Ma'aita, Assistant Professor - Consultant endodontist, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10/2017/25289
Record Dates: First submitted 2018-04-01; First posted 2018-05-31 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pulp Disease, Dental; Dental Caries; Dental Leakage
MeSH Terms: conditions — Dental Pulp Diseases; Dental Caries; Dental Leakage | interventions — Dental Prosthesis; Crowns

STUDY DESIGN:
Intervention Model Description: Three different ceramic types for restoration of endodontically treated teeth
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All ceramic materials will be assigned randomly by research assistant who has randomised tables generated by a statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lithium disilicate (Active Comparator): Lithium disilicate: a type of ceramic material used to make a dental prosthesis that replaces missing tooth structure following root canal treatment. Other names might include: E-max crowns, computer-aided design and computer-aided manufacturing (CAD CAM) crowns
  Interventions: Device: Dental prosthesis
- Monolithic zirconia (Active Comparator): Monolithic zirconia: a type of ceramic material used to make a dental prosthesis that replaces the missing tooth structure following root canal treatment. Other names might include: Zolid crown, Bruxzir, Bretau, CAD CAM crowns
  Interventions: Device: Dental crown
- Hybrid ceramic (Active Comparator): Hybrid ceramic: a type of ceramic material used to make a dental prosthesis that replaces the missing tooth structure following root canal treatment. Other names might include: Enamec, Lava Ultimate, CAD CAM crowns
  Interventions: Device: Hybrid ceramic

INTERVENTIONS:
Device: Dental prosthesis — Replacement of missing tooth structure using Lithium disilicate porcelain
  Other Names: Crowns
  Arms: Lithium disilicate
Device: Dental crown — Replacement og missing tooth structure using monolithic zirconia
  Other Names: Endocrown
  Arms: Monolithic zirconia
Device: Hybrid ceramic — Restroration of endodontically treated teeth using hybrid ceramic
  Other Names: Indirect restoration
  Arms: Hybrid ceramic

SUMMARY:
Restoration of endodontically treated teeth requires a means to protect the cusps from the wedging forces of occlusion. When there is extensive loss of tooth structure, cuspal coverage is warranted. Usually this is in the form of indirect restoration. Traditionally, full coverage crowns have been used which would require further removal of sound tooth structure. Recently, adhesive alternatives have been introduced which allow for conservation of tooth structure.

Different materials can be used for this purpose. The evidence on the long-term survival of these materials is scarce. This study aims to investigate the short and medium-long term survival rate of these prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Root canal treated molars with significant loss of tooth structure
* Supra-gingival margins
* Teeth scheduled for cuspal-covering indirect restorations

Exclusion Criteria:

* Teeth with extensive cracks or fractures
* Teeth with deep subgingival margins
* Non-functional teeth (no opposing dentition)
* Teeth with advanced periodontitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lithium Disilicate | Monolithic Zirconia | Hybrid Ceramic
Started | 20 | 20 | 20
Completed | 19 | 17 | 19
Not Completed | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium Disilicate | Monolithic Zirconia | Hybrid Ceramic | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (10.6) | 38.1 (14.9) | 33.4 (11.2) | 34.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 11 | 39
  Male | 5 | 7 | 9 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Jordan | 20 | 20 | 20 | 20

OUTCOME MEASURES:

1. Primary Outcome: Survival of Dental Prosthesis
Description: The endocrowns (the dental prosthesis studied) were assessed after 24 months. Those that were functional and without any symptoms were considered surviving.
Time Frame: 24 months
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Lithium Disilicate | Monolithic Zirconia | Hybrid Ceramic
Number analyzed (Participants) | 16 | 17 | 18
Number analyzed (Teeth) | 19 | 17 | 19
Teeth | 19 | 14 | 17

ADVERSE EVENTS:
Time Frame: 24 months
Description: Debonding, fracture, poor appearance, or if the tooth was deemed non-restorable during the 24-month observation period.
Arm/Group | Lithium Disilicate | Monolithic Zirconia | Hybrid Ceramic
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 3/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Disilicate (N=20) | Monolithic Zirconia (N=20) | Hybrid Ceramic (N=20)
Debonding (Product Issues) | 0 (0) | 3 (3) | 2 (2) — Endocrown/ dental prosthesis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT03542019/Prot_SAP_000.pdf